CLINICAL TRIAL: NCT00526760
Title: A Phase 3, Open-Label Study Evaluating the Safety and Efficacy of Dexmedetomidine in ICU Subjects Requiring Greater Than 24 Hours of Continuous Sedation
Brief Title: Long-term Clinical Study Evaluating the Safety and Efficacy of Dexmedetomidine in ICU Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Maruishi Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEX-402
Record Dates: First submitted 2007-09-05; First posted 2007-09-10 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Sedation
Keywords: Dexmedetomidine, Sedation, Long-term, Phase 3
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine

SUMMARY:
Evaluate efficacy and safety of dexmedetomidine long term administration in ICU patients who require more than 24 hours sedation.

DETAILED DESCRIPTION:
According to the current dexmedetomidine indication, the duration of dexmedetomidine administration is limited within 24 hours. However, there is a strong demand from the medical specialists for continued administration of dexmedetomidine in excess of 24 hours in the medical practice because a large number of patients require sedation for more than 24 hours in ICU. To meet such clinical demand, it was planned to conduct a phase III long-term administration study of dexmedetomidine to obtain the approval on the infusion of dexmedetomidine for more than 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or legally acceptable representative (if acceptable by Institutional Review Board/Ethics Committee) has signed and dated the Informed Consent after the study had been fully explained.
2. Patient is male or female, at least 20 years of age.
3. In case of surgical ICU patient, who is in condition of American Society of Anesthesiologists (ASA) I to III Class preoperatively.
4. Patient is on mechanical ventilation and anticipated to require sedation more than 24 hours following a surgery.
5. If patient is female with child bearing potential, she is to be non-pregnant, and not lactating.

Exclusion Criteria:

1. Patient has serious central nervous system (CNS) trauma.
2. Patient requires the use of neuromuscular blocking agents after admission to ICU, except for the insertion of the endotracheal tube.
3. Patient is hospitalized for drug overdose within the last 30 days.
4. Patient in whom alpha-2 antagonists or alpha-2 agonists are contraindicated.
5. Patient is currently being treated or has been treated within the last 30 days with alpha-2 agonist or antagonist.
6. Patient has participated in a trial with any experimental drug within 30 days prior to admission to the ICU.
7. Terminally ill patient, whose life duration expectancy is no more or around 30 days.
8. Patient is considered unable to undergo any procedure required by the protocol.
9. Patient with excessive bleeding which will likely require surgery.
10. In the Investigator's opinion, patient has any symptom or factor, which might increase risk to the patient or preclude obtaining satisfactory study data.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Incidence rate of adverse drug reactions of hypotension, hypertension and bradycardia which correspond to the protocol definitions | Prior to study drug infusion, during the study drug infusion and 24 hours after study drug infusion end; maximum ≤28 days.
  Definition:
  * Hypotension: dosing start or dose increase of vasopressor drug or use of fluid bolus ≥500 mL within 1 hour resulting from SBP<60mmHg, DBP<40mmHg or ≥50% lower than baseline.
  * Hypertension: dosing start or dose increase of intravenous anti-hypertensive medication resulting from SBP>160, DBP>100 or. ≥50% higher than baseline.
  * Bradycardia: dosing start or dose increase of positive chronotropic medication or use of pacemaker resulting from heart rate <40bpm or ≥50% lower than baseline.

SECONDARY OUTCOMES:
Percentage of with a Richmond Agitation-Sedation Sedation Score ≤0 during the study drug infusion | Prior to study drug infusion, during the study drug infusion and 24 hours after study drug infusion end; maximum ≤28 days.
Percentage of time with a Richmond Agitation-Sedation Sedation Score =0, -1,-2 during the study drug infusion | Prior to study drug infusion, during the study drug infusion and 24 hours after study drug infusion end; maximum ≤28 days.
Administration frequency and dosage of additional sedatives | Prior to study drug infusion, during the study drug infusion and 24 hours after study drug infusion end; maximum ≤28 days.
Administration frequency and dosage of additional analgesics | Prior to study drug infusion, during the study drug infusion and 24 hours after study drug infusion end; maximum ≤28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Misa Kawai, Study Director — Hospira, now a wholly owned subsidiary of Pfizer
Locations (10):
- Japan (10):
  - Hyogo Medical University Hospital, Nishinomiya, Hyōgo
  - Kagoshima University Hospital, Kagoshima, Kagoshima-ken
  - Kinki University Hospital, Sayama, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Hamamatsu Medical University Hospital, Hamamatsu, Shizuoka
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - Jikei University Hospital, Minato-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - Keio University Hospital, Sinjuku-ku, Tokyo
  - Yamanashi University Hospital, Chūō, Yamanashi